CLINICAL TRIAL: NCT04290715
Title: Development and Validation for Predicting Inadequate Bowel Preparation Before Colonoscopy in Patients
Brief Title: Development and Validation for Predicting Inadequate Bowel Preparation
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IBPN-V1.0
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Polyethylene Glycol; Cathartics; Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A
  Interventions: Other: no intervention
- group I
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
High-quality colonoscopy is considered the gold standard for the detection and prevention of colorectal cancer, and its efficacy is predicated on optimal colon cleansing.However, about 18%-35% of patients were still reported to suffer inadequate bowel preparation. Although several predictive models exist, the current guideline indicates that there is insufficient evidence to recommend the use of a predictive model for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing colonoscopy.
* patients older than 18 years.

Exclusion Criteria:

* Emergency colonoscopy.
* Have a serious medical condition, such as heart failure, acute liver failure, severe kidney disease (dialysis or predialysis patients) or New York heart association class iii-iv.
* Pregnant or breastfeeding.
* No bowel preparation or poor compliance (no bowel preparation as instructed or laxatives < 90% of prescribed dose).
* Refuse to sign informed consent.
* The patient was rescheduled after the previous colonoscopy due to insufficient bowel preparation.
* Temporarily change to colonoscopy for other reasons.
* Incomplete colonoscopy due to insufficient parenteral preparation.
* Lack of complete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. patients undergoing colonoscopy.
  2. patients older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1644 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
quality of bowel preparation | A colonoscopy procedure
  The OBPS is a validated scoring system with scores between 0 and 14, where 0 is the best score. The score comprises a sub score 0-4 for each colon segment: right, transverse and rectosigmoid colon. In addition, a score 0-2 is added to indicate the total amount of luminal fluid.
  For all participants, OBPS score will be used when the colonscopy is inserting.
quality of bowel preparation | A colonoscopy procedure
  The BBPS is another validated scoring system with scores between 0 and 9, where 9 is the best score. The score comprises a sub score 0-3 for each colon segment: right, transverse and left colon.
  For all participants, BBPS score will be used when colonscopy is withdrawing.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China